CLINICAL TRIAL: NCT04703517
Title: Musculoskeletal Ultrasonography to Diagnose Successful Reduction of Shoulder Dislocation
Brief Title: Musculoskeletal Ultrasound for Diagnosis of Shoulder Dislocation Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Jesper Aurup, MD, MD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro2020003069
Record Dates: First submitted 2020-12-16; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Ultrasound; Shoulder Dislocation; Musculoskeletal Injury
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self Controlled (Other): Patients will active as their own comparator
  Interventions: Diagnostic Test: Point of care ultrasound

INTERVENTIONS:
Diagnostic Test: Point of care ultrasound — Patients will receive a point of care ultrasound at the bedside in the Emergency Department and compare the impression to the x ray result

SUMMARY:
This study will compare the current standard of care post reduction plain film x ray for confirmation of shoulder reduction to point of care ultrasound. Patients will receive both the current standard of care post reduction x ray and point of care ultrasound to act as their own comparators

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to 18 years
* Acute shoulder dislocation

Exclusion Criteria:

* Associated fracture
* Associated neurovascular injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of X ray to Ultrasound for Shoulder Reduction | through study completion up to 1 year
  Compare the impression of the x ray to the ultrasound for successful shoulder reduction

SECONDARY OUTCOMES:
Comparison of X ray to Ultrasound in the diagnosis of post shoulder reduction complications | through study completion up to 1 year
  Compare the impression of the x ray to the ultrasound for shoulder dislocation complications

IPD SHARING:
Plan to Share IPD: No